CLINICAL TRIAL: NCT05041205
Title: Functional Test for a Drink Powder: a Randomized, Double-blind, Placebo-controlled Human Consumption Test
Brief Title: Functional Test for a Drink Powder Alone and Combined Use With a Cosmetic Apparatus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C210201
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Beauty Drink Powder; Cosmetic Apparatus on Skin; Skin Elasticity; Skin Dryness; Skin Moisture; Skin Evenness; Skin Firmness

STUDY DESIGN:
Intervention Model Description: Participants are assigned to four group during the study: a placebo control group, a beauty drink powder group, a cosmetic apparatus group, and a beauty drink powder + cosmetic apparatus group
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, participants and outcomes assessors are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo control group (Placebo Comparator): placebo drink powder without active ingredients, 1 sachet per day with 50 ml water for 12 weeks
  Interventions: Dietary Supplement: Beauty drink powder
- Beauty drink powder group (Experimental): Beauty drink powder is the test article provide to participants, 1 sachet per day with 50 ml water for 12 weeks
  Interventions: Dietary Supplement: Beauty drink powder
- cosmetic apparatus group (Placebo Comparator): This group is designed for a cosmetic apparatus control group without consumption of placebo or test article. Together with the specified cleanser, the apparatus is used for daily facial cleaning, two times in the morning and evening for 12 weeks.
  Interventions: Device: Cosmetic apparatus
- Beauty drink powder + cosmetic apparatus group (Experimental): In this group, Beauty drink powder is consumed 1 sachet daily with 50 ml water and the cosmetic apparatus is used together with the specified cleanser for daily facial cleaning, two times in the morning and evening for 12 weeks.
  Interventions: Dietary Supplement: Beauty drink powder; Device: Cosmetic apparatus

INTERVENTIONS:
Dietary Supplement: Beauty drink powder — Beauty drink powder is designed as a oral beauty product to provide benefits to skin
  Arms: Beauty drink powder + cosmetic apparatus group; Beauty drink powder group; Placebo control group
Device: Cosmetic apparatus — This device is designed to let participants to experience brighter, softer, smoother skin and an energizing facial massage. A synergestic effect when combine with beauty drink powder is expected.
  Arms: Beauty drink powder + cosmetic apparatus group; cosmetic apparatus group

SUMMARY:
This study is designed to observe human consuming effect of a beauty drink powder and combined use with a cosmetic apparatus. It is a randomized, double-blind, and placebo-control study. The target enrollment of subjects is 160 and 4 arms are included, a placebo control, drink powder alone, cosmetic apparatus alone, and drink powder plus cosmetic apparatus. Effects on skin dullness, skin tone unevenness, skin dryness, skin elasticity, wrinkle and fine line are evaluated. Both objective and subjective methods are used for efficacy evaluation. Data are collected at baseline, week 4, week 8, and week 12 after treatment.

DETAILED DESCRIPTION:
In this study, objective parameters are measured by the instruments as following: VisioScan VC20 is used for skin roughness and wrinkle assessment, chromameter CR-400 is used to assess skin color, skin gloss is assessed by Glossymeter, skin hydration is assessed by Corneometer, TEWL is assessed by Vapometer, and skin elasticity is assessed by Cutometer. VISIA-CR and VISIA-7 are used in skin radiation and wrinkle visualization.

Clinical assessment is performed by expert visual grading on

* Skin evenness
* Skin radiance
* Skin elasticity
* Skin smoothness
* Skin firmness
* Skin moisture
* Skin plumpness

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male or female
* Subjects with skin problems such as skin dullness, skin tone unevenness, skin inelasticity, skin dryness, and wrinkle/fine lines.
* Subjects without any other chronic or on treatment diseases
* Subjects are voluntary to participate the trial and signed informed consents.
* Subjects are voluntary to follow all evaluation criteria

Exclusion Criteria:

* Subjects have a plan to be pregnant, or are in pregnancy or lactation period;
* Not participated any clinical trial or evaluation within nearly 1 month;
* Used anti-histamine medication within nearly one week or immunosuppressor within nearly one month
* Used any anti-inflammation drugs at test site within nearly two months
* Subjects who have any skin diseases (psoriasis, eczema, skin cancer etc.)
* Subjects with Type I diabetes
* Subjects who currently are receiving asthma or other chronic respiratory diseases treatment
* Subjects who are receiving anti-cancer chemotherapy in nearly 6 months
* Subjects who have anyother health problem or chronic diseases
* Subjects who have externally used Vit A, a-hydroxy acid, salicylic acid, hydroquinone within nearly 3 months or prescription medicines, oral contraceptive within nearly 6 months
* Expert or professional person evaluate have other iatrogenic reason may impact the evaluation results

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Skin health (evenness) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of evenness (using scores from 0-10 to indicate skin evenness from evenness to unevenness) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (radiance) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of radiance (using scores from 0-10 to indicate skin radiance from radiance to dulness) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (elastisity) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of elastisity (using scores from 0-10 to indicate skin elasticity from elastic to nonelastic) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (smoothness) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of smoothness (using scores from 0-10 to indicate skin smoothness from smooth to rough) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (firmness) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of firmness (using scores from 0-10 to indicate skin firmness from firm to slack) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (moisture) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of moisture (using scores from 0-10 to indicate skin moisture from moist to dry) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (plumpness) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of plumness (using scores from 0-10 to indicate skin plumpness from plump to not plump) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data
Skin health (overall) | baseline, day 28, day 56, and day 84
  Change from baseline in investigator facial grading of overall (using scores from 0-10 to indicate overall skin health from good to worse) at days 28, 56, and 84 using Wilcoxon and Mann Whitney two tailed assessment for nonparametric data

SECONDARY OUTCOMES:
Skin roughness and wrinkle of face determined by VisioScan VC20 | Baseline, day 28, day 56, and day 84
  Change from baseline in skin roughness and wrinkle at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data
Skin Color of L, a, b and ITA value of face determined by chromameter | Baseline, day 28, day 56, and day 84
  Change from baseline in skin color of L, a, b, and ITA value at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data
Skin Glossiness of face determined by Glossymeter | Baseline, day 28, day 56, and day 84
  Change from baseline in skin glossiness at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data
Skin hydration of face determined by Corneometer | Baseline, day 28, day 56, and day 84
  Change from baseline in skin hydration at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data
Face TEWL determined by Vapometer | Baseline, day 28, day 56, and day 84
  Change from baseline in face TEWL at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data
Skin elasticity of face determined by Cutometer | Baseline, day 28, day 56, and day 84
  Change from baseline in skin elasticity at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data
Skin radiance and lines assessed by facial photo capture using VISIA-CR and VISIA-7 | Baseline, day 28, day 56, and day 84
  Change from baseline in skin radiance and lines at days 28, 56, and 84 using Wilcoxon and Mann-Whitney test for nonparametric data

CONTACTS AND LOCATIONS:
Overall Officials: Wenwen Gu, PhD, Principal Investigator — Shanghai China-norm Quality Technical Service Co., Ltd.
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No